CLINICAL TRIAL: NCT02823743
Title: Treatment of Recurrent Abortion With Low Dose Aspirin - a Randomized Placebo Controlled Trial
Brief Title: RECAB-ASA; Treatment of Recurrent Abortion With Aspirin
Acronym: RECAB-ASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Annika Strandell, Associate professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGR-2170
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Abortion, Habitual
Keywords: recurrent pregnancy loss, Habitual abortion
MeSH Terms: conditions — Abortion, Habitual | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose aspirin (Experimental): 75 mg aspirin orally daily from gestational week 7-35
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo pill orally daily from gestational week 7-35
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Daily medication
  Other Names: ASA
  Arms: Low dose aspirin
Drug: Placebo — Daily intake
  Arms: Placebo

SUMMARY:
The aim of this study is to examine whether treatment with 75 mg aspirin daily compared with placebo could reduce the risk for a new miscarriage. The treatment starts when the pregnancy is detected on transvaginal ultrasound (around gestational week 6+) and continues to week 35/36. The study is a single center, randomized, placebo-controlled, double blind and stratified for age. 400 participants with the diagnosis idiopathic recurrent abortion are enrolled, 200 in each arm aspirin / placebo.

ELIGIBILITY:
Inclusion Criteria:

* recurrent abortion (≤ 3 consecutive abortions in first trimester)
* unknown etiology after work-up
* willingness to be randomized

Exclusion Criteria:

* previous participation in the study
* known cause of recurrent abortion, requiring specific management
* age ≥ 40
* BMI above 35
* IVF pregnancy if the reason for IVF was recurrent spontaneous abortion
* ongoing treatment with aspirin for other reason
* Sjoegren syndrome

Max Age: 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2008-03; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Live birth | delivery

SECONDARY OUTCOMES:
Spontaneous abortion | up to 22 weeks
Vaginal bleeding | up to 42 weeks
Premature delivery | At delivery
intrauterine growth retardation, measured by ultrasound as percentage deviation | up to 42 weeks
Preeclampsia | up to 42 weeks
Pregnancy induced hypertension | up to 42 weeks
Placenta praevia | up to 42 weeks
Perinatal mortality | Third trimester and 28 days after delivery
Perinatal morbidity | 28 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Annika Strandell, Ass.prof., Principal Investigator — Göteborg University

IPD SHARING:
Plan to Share IPD: Undecided